CLINICAL TRIAL: NCT06550466
Title: The Influence of Pre-exercise Feeding on Acute Bone Turnover Biomarkers in Response to Physical Activity in Healthy Participants
Brief Title: The Effect of Pre-exercise Feeding on Bone Turnover Biomarkers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Anglia Ruskin University (Other); University of Sheffield (Other); Manchester Metropolitan University (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ER52048815
Record Dates: First submitted 2024-07-30; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Osteopenia or Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis

STUDY DESIGN:
Intervention Model Description: In this three-arm randomised crossover study, sixteen young adult men (age: 28 ± 4) will be recruited in good physical condition. Participants will be exercised following a 12-hour overnight fast (FAST) and exercised 90 minutes after a meal (FED) to test the temporal sensitivity of the loaded bone to absorbed nutrients. Participants will also attend a breakfast-only arm (without the exercise protocol).
  Participants will undergo a baseline assessment for health history (PAR-Q). The blood samples will be collected (10ml) and osteogenic response to exercise will be determined by measuring markers of bone formation; P1NP and resorption; CTX-1 and cortisol; marker of physiological and psychological stress. Insulin and glucose measurements will allow to assess the change of concentrations in fasted and fed states.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breakfast only (Experimental): Breakfast only without the exercise protocol
  Interventions: Other: Breakfast only
- FAST (Experimental): Participants will be exercised 90 minutes following a 12-hour overnight fast
  Interventions: Other: FAST
- FED (Experimental): Participants will be exercised 90 minutes after a meal
  Interventions: Other: FED

INTERVENTIONS:
Other: Breakfast only — Participants will attend a breakfast-only arm without the exercise protocol.
  Arms: Breakfast only
Other: FAST — Participants will be exercised for 90 minutes following a 12-hour overnight fast
  Arms: FAST
Other: FED — Participants will be exercised 90 minutes after a breakfast
  Arms: FED

SUMMARY:
Osteoporosis is a major contributor to loss of independence due to bone fractures and resulting hospital treatments lead to significant morbidity. While pharmacological treatments can reduce consequences of osteoporosis, there is a pressing need for non-pharmacological interventions to improve bone health across the life-course and to reduce likelihood of age-related bone disease.

This study will allow us to determine whether synergistic potentiating effects on bone metabolism are observed in humans in relation to the timing of food ingestion and what recommendations can be made to people with respect to food ingestion and exercise to obtain the maximal bone benefits from aerobic exercise. Furthermore, if we can identify interventions that potentiate bone's response to aerobic exercise in younger adults, then such interventions may have the ability to maximise bone mass in younger adults so that with ageing, the additional bone mineral density and improved bone microarchitecture would extend the time before osteoporotic "fracture thresholds" are reached. Therefore, understanding the bone metabolic response to exercise following fasting and feeding in younger adults is important.

ELIGIBILITY:
Inclusion Criteria:

* Male (females excluded to remove the interplay between menstrual cycle and bone turnover)
* Caucasian ethnicity
* Aged 28 ± 4 years
* Are physically active (meet the UK guidelines for physical activity of at least 150 minutes moderate intensity activity and/or at least 75 minutes of vigorous intensity activity per week)
* Otherwise, healthy, able and willing to participate and provide written informed consent

Exclusion Criteria:

* Current smokers
* Excessive alcohol consumption (max 15 alcohol units/week)
* Any musculoskeletal injury/disabilities
* Any conditions known to affect bone metabolism (e.g. uncontrolled hyper-/hypothyroidism, hyperparathyroidism, hypo-/hypercalcaemia) or malabsorption syndromes (e.g. Crohn's disease, coeliac disease or inflammatory bowel disease).
* Taking any medication known to affect bone metabolism (such as glucocorticoids or bisphosphonates)
* Positive Covid-19 test within the last 8 weeks
* Suffered a fracture in the previous 12 months
* Sedentary status (see physical activity inclusion criteria above)
* Have been told by medical professionals that they should not take part in moderate to high intensity exercise
* Should not be a professional athlete or take part in significant competitive recreational activity (takes no more than 4 structured exercise sessions per week on average)
* History of diagnosed eating disorders

Ages: 24 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
C-terminal telopeptide of type-1 collagen (CTX-1) | Between pre-exercise and 2 hours following the exercise timepoints
  The primary endpoint of this study is the change of the bone resorption biomarker C-terminal telopeptide of type-1 collagen (CTX-1) expression

SECONDARY OUTCOMES:
Procollagen type 1 N-terminal propeptide (P1NP) | Between pre-exercise and 2 hours following the exercise timepoints
  The change of the bone formation biomarker procollagen type 1 N-terminal propeptide (P1NP) expression
Cortisol | Between pre-exercise and 2 hours following the exercise timepoints
  Markerof physiological and psychological stress is assessed and because of its promotion of bone resorption
Insulin | Between pre-exercise and 2 hours following the exercise timepoints
  The change of concentration in fasted and fed states is assessed
Glucose | Between pre-exercise and 2 hours following the exercise timepoints
  The change of concentration in fasted and fed states is assessed

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-30): https://cdn.clinicaltrials.gov/large-docs/66/NCT06550466/Prot_SAP_000.pdf